CLINICAL TRIAL: NCT00083213
Title: An Open Label, Sequential Cohort Dose-Escalation Safety, Tolerability and Pharmacokinetic Study of VEGF Trap Administered Intravenously in Patients With Advanced Solid Tumors or Lymphoma
Brief Title: Intravenous VEGF Trap in Treating Patients With Relapsed or Refractory Advanced Solid Tumors or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REGENERON-VGFT-ST-0202; MSKCC-03137; CDR0000360856 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Cancer
Keywords: recurrent grade 1 follicular lymphoma; stage IV grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; stage IV grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; recurrent adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; recurrent adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; recurrent mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; unspecified adult solid tumor, protocol specific; recurrent adult soft tissue sarcoma; recurrent adult primary liver cancer; advanced adult primary liver cancer; recurrent cervical cancer; stage IVA cervical cancer; stage IVB cervical cancer; fallopian tube cancer; ovarian sarcoma; recurrent ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent endometrial carcinoma; stage IV endometrial carcinoma; recurrent uterine sarcoma; stage IV uterine sarcoma; recurrent ovarian germ cell tumor; stage IV ovarian germ cell tumor; ovarian stromal cancer; recurrent vaginal cancer; stage IVA vaginal cancer; stage IVB vaginal cancer; recurrent prostate cancer; stage IV prostate cancer; recurrent penile cancer; stage IV penile cancer; recurrent malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; recurrent bladder cancer; stage IV bladder cancer; recurrent vulvar cancer; stage IVB vulvar cancer; distal urethral cancer; proximal urethral cancer; recurrent urethral cancer; urethral cancer associated with invasive bladder cancer; primary peritoneal cavity cancer; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Neoplasms; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Sarcoma; Carcinoma, Hepatocellular; Uterine Cervical Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial; Endometrial Neoplasms; Vaginal Neoplasms; Prostatic Neoplasms; Penile Neoplasms; Testicular Neoplasms; Urinary Bladder Neoplasms; Vulvar Neoplasms; Urethral Neoplasms; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — aflibercept

INTERVENTIONS:
Biological: ziv-aflibercept

SUMMARY:
RATIONALE: VEGF Trap may stop the growth of solid tumors or non-Hodgkin's lymphoma by stopping blood flow to the tumor.

PURPOSE: This phase I trial is studying the side effects and best dose of intravenous VEGF Trap in treating patients with relapsed or refractory advanced solid tumors or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and tolerability of intravenous VEGF Trap in patients with relapsed or refractory advanced solid tumors or non-Hodgkin's lymphoma.

Secondary

* Determine the maximum tolerated intravenous dose of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Determine the ability of this drug to bind circulating vascular endothelial growth factor in these patients.
* Determine, preliminarily, the ability of this drug to alter tumor blood flow and tumor vascular permeability in these patients.
* Determine whether antibodies to this drug develop in these patients.

OUTLINE: This is an open-label, dose-escalation, multicenter study.

Patients receive VEGF Trap IV over 1 hour on days 1 and 15 for a total of 2 doses.

Cohorts of 3-6 patients receive escalating doses of VEGF Trap until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional 6 patients are treated at that dose level.

In the absence of dose-limiting toxicity, patients with stable disease or partial or complete remission may continue to receive VEGF Trap on a separate extension protocol.

Patients are followed at weeks 1, 3, and 7 and then at 3 months.

PROJECTED ACCRUAL: A maximum of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of one of the following:

  * Non-Hodgkin's lymphoma
  * Primary or metastatic solid tumor located, by radiography, in at least one of the following sites:

    * Liver
    * Soft tissue
    * Pelvis
    * Other site that is suitable for delayed contrast-enhanced MRI (e.g., peripheral lung field)
* Relapsed or refractory (including unresectable) disease

  * Patients with solid tumors must have failed all curative chemotherapeutic regimens
  * Patients with non-Hodgkin's lymphoma must be refractory to at least 2 standard chemotherapeutic regimens and rituximab
* Not amenable to available conventional therapies AND no standard therapy exists
* Measurable disease
* No prior or concurrent CNS metastases (brain or leptomeningeal)
* No primary intracranial tumor by MRI or CT scan
* No histologically confirmed squamous cell carcinoma of the lung

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,500/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100,000/mm^3
* No severe or uncontrolled hematologic condition

Hepatic

* Bilirubin ≤1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* PT and PTT normal
* INR normal
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal

* Creatinine ≤ ULN
* Urine protein/creatinine ratio ≤ 1
* No severe or uncontrolled renal condition

Cardiovascular

* No clinically significant acute electrocardiographic abnormalities
* LVEF normal by echocardiogram or MUGA within the past 12 months if there was prior exposure to anthracyclines
* No untreated or uncontrolled hypertension

  * No blood pressure > 150/100 mm Hg (despite treatment)
* No isolated systolic hypertension (i.e., systolic blood pressure > 180 mm Hg on at least 2 determinations [on separate days] within the past 3 months)
* No New York Heart Association class II - IV heart disease
* No active coronary artery disease requiring acute medical management
* No angina requiring acute medical management
* No congestive heart failure requiring acute medical management
* No ventricular arrhythmia requiring acute medical management
* No stroke or transient ischemic event within the past 6 months
* No prior or concurrent peripheral vascular disease

  * No angiographically or ultrasonographically documented arterial or venous occlusive event
  * No symptomatic claudication
* No symptomatic orthostatic hypotension
* No other severe or uncontrolled cardiovascular condition

Pulmonary

* No severe or uncontrolled pulmonary condition
* No pulmonary embolism within the past 6 months

Immunologic

* HIV negative
* No severe or uncontrolled immunologic condition
* No active current infection requiring antibiotics
* No prior hypersensitivity reaction to any recombinant proteins, including VEGF Trap

Other

* No severe or uncontrolled gastrointestinal or musculoskeletal condition
* No psychiatric condition or adverse social circumstance that would preclude study participation
* No other condition that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-barrier contraception during and for 3 months after study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior participation in a VEGF Trap, interleukin-1 Trap, or interleukin-4/13 Trap clinical trial
* At least 3 weeks since prior immunotherapy and recovered
* No concurrent epoetin alfa, filgrastim (G-CSF), or sargramostim (GM-CSF)

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy and recovered

Endocrine therapy

* No concurrent adrenal corticosteroids except low-dose replacement therapy
* No concurrent systemic hormonal contraceptive agents

Radiotherapy

* At least 3 weeks since prior radiotherapy and recovered

Surgery

* At least 3 weeks since prior major or laparoscopic surgery and recovered
* More than 6 months since prior surgical procedure for correction or prophylaxis of peripheral vascular insufficiency or cerebral ischemic events

Other

* More than 30 days since prior investigational drugs
* No concurrent anticoagulant or antiplatelet drugs (e.g., warfarin, heparin, or aspirin) other than low-dose (1 mg) warfarin for maintaining patency of venous access devices
* No concurrent non-steroidal anti-inflammatory drugs, including cyclo-oxygenase-2 (COX-2) inhibitors
* No other concurrent anticancer investigational agents
* No other concurrent anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-01; Primary Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William P. Tew, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan - Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Lockhart AC, Rothenberg ML, Dupont J, Cooper W, Chevalier P, Sternas L, Buzenet G, Koehler E, Sosman JA, Schwartz LH, Gultekin DH, Koutcher JA, Donnelly EF, Andal R, Dancy I, Spriggs DR, Tew WP. Phase I study of intravenous vascular endothelial growth factor trap, aflibercept, in patients with advanced solid tumors. J Clin Oncol. 2010 Jan 10;28(2):207-14. doi: 10.1200/JCO.2009.22.9237. Epub 2009 Nov 30. PMID 19949018
- [Result] Wang-Gillam A, Tew WP, Rothenberg ML, Dupont J, Cooper W, Sternas L, Buzenet G, Sosman JA, Spriggs DR, Lockhart AC. A phase I study of subcutaneously administered aflibercept (VEGF trap) in a new formulation in patients with advanced solid tumors. Invest New Drugs. 2012 Oct;30(5):1958-61. doi: 10.1007/s10637-011-9753-y. Epub 2011 Oct 15. PMID 22002018